CLINICAL TRIAL: NCT04628559
Title: Comparison of the Perioperative Effects of Dexmedetomidine and Ketamine Sedation in Septorhinoplasty Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Muge Kosucu, Clinical Associated Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009/137
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Anesthesia; Intravenous Anesthetic Toxicity
Keywords: Dexmedetomidine; Ketamine; Perioperative effects
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 1. First arm received dexmedetomidine
  2. Second arm received ketamine
  3. Third arm received saline solution.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The surgeon and observers were all blinded to the patients until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomine (Active Comparator): Patients recieving Dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- Ketamine (Active Comparator): Patients recieving Ketamine.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Patients recieving Saline.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine was administered as a gradual bolus of 1 µg/kg/10ml 10 min before induction of anesthesia and then as an infusion of 0.4 µg/kg per min (30 ml/h). In Group K, ketamine was administered as a 0.4 mg/kg/10ml IV bolus 10 min before induction of anesthesia and in the form of 10 µg/kg per min infusion after induction (30 ml/h).
  Other Names: Group D
  Arms: Dexmedetomine
Drug: Ketamine — In Group K, ketamine was administered as a 0.4 mg/kg/10ml IV bolus 10 min before induction of anesthesia and in the form of 10 µg/kg per min infusion after induction (30 ml/h).
  Other Names: Group K
  Arms: Ketamine
Drug: Saline — Group S was given a bolus of saline solution in 10 ml volume 10 min before induction of anesthesia, followed by 30 mL/h serum saline infusion.
  Other Names: Group S
  Arms: Placebo

SUMMARY:
This randomized double-blind study aimed to compare the effects of dexmedetomidine and ketamine on hemodynamic parameters, recovery criteria, and opioid consumption and advers effects in septorhinoplasty operations. Totally 63 patients were included.

The groups were compared in terms of hemodynamic values, recovery times, postoperative agitation, sedation, activity, modified Aldrete and pain scores, side-effects and additional analgesia requirements at postoperative 24h.

DETAILED DESCRIPTION:
A total of 63 patients 18-55 years undergoing septorhinoplasty, who were graded as American Society of Anesthesiologists physical status were randomly allocated into three groups, receiving dexmedetomidine (n=21, Group D), ketamine (n=21, Group K) and saline solution (n=21, Group S). Anesthesia was induced with propofol, cisatracurium and fentanyl. Maintenance anesthesia was done with 2-2.5% sevoflurane mixture, 50-60% oxygen and N2O. The groups were compared in terms of hemodynamic values, recovery times, postoperative agitation, sedation, activity, modified Aldrete and pain scores, side-effects and additional analgesia requirements at postoperative 24h.

ELIGIBILITY:
Inclusion Criteria:

* Patient graded as American Society of Anesthesiologist (ASA) physical status, I or II
* Patient subjected to septorhineoplasty operation

Exclusion Criteria:

* Patient having morbid obesity,
* Patient having yypertension,
* Patient having Asthma,
* Patient having neuropsychiatric disease,
* Patient allergy to the study drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2009-12-30 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Response to verbal stimulus time | 0-120 minutes following finishing operation
  Verbal response received when the patient was spoken to
Intraoperative additional fentanyl requirement | 0-120 minutes following initiating operation
  Intraoperative additional fentanyl requirement for pain relief and

SECONDARY OUTCOMES:
Heart rate | 0-120 minutes
  Heart rate during operation and following operation

CONTACTS AND LOCATIONS:
Overall Officials: Muge Muge, Assoc Prof, Study Chair — Medical School of Karadeniz Technical University, Department of Anesthesiology
Locations (1):
- Medical School of Karadeniz Technical University, Department of Anesthesiology, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No